CLINICAL TRIAL: NCT06553027
Title: Phase 3, Randomized, Double-Blind, Placebo-Controlled Multicenter Study of CVN424 in Parkinson's Disease Patients With Motor Complications
Brief Title: To Evaluate the Efficacy of CVN424 in Parkinson's Disease Participants With Motor Complications
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cerevance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVN424-301; 2024-516811-25-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-09; First posted 2024-08-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; CVN424; Phase 3; Motor fluctuations; Idiopathic Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CVN424 75 mg (Experimental): Participants will be administered with oral doses of 75 mg CVN424.
  Interventions: Drug: CVN424 75 mg
- CVN424 150 mg (Experimental): Participants will be administered with oral doses of 150 mg CVN424.
  Interventions: Drug: CVN424 150 mg
- Placebo (Placebo Comparator): Participants will be administered with placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CVN424 75 mg — Participants will receive 75 mg CVN424 tablet once daily.
  Arms: CVN424 75 mg
Drug: CVN424 150 mg — Participants will receive 150 mg CVN424 tablet once daily.
  Arms: CVN424 150 mg
Drug: Placebo — Participants will receive matching placebo tablet once daily.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter study in participants with Parkinson's disease (PD) with motor fluctuations. Participants will be randomized to receive once-daily oral doses of either 75 milligrams (mg) CVN424 or 150 mg CVN424, or a matching placebo for 12 weeks. Participants who successfully complete this study and retain eligibility/suitability will be invited to participate in a future open-label extension (OLE) study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD consistent with United Kingdom (UK) Brain Bank criteria and MDS Research Criteria for the Diagnosis of PD; must include bradykinesia with sequence effect and motor asymmetry if no rest tremor, and a prominent response to levodopa.
* Body Mass Index (BMI) > 18.0 and < 35.0 Kilograms per meter square (kg/m^2), inclusive at Screening.
* Modified Hoehn and Yahr Stage ≤ 3 in the ON state.
* Freely ambulatory at the time of Screening (with/without assistive device).
* Montreal Cognitive Assessment (MoCA) Score of at least 24.
* PD medications must be stable for at least 4 weeks prior to Screening; monoamine oxidase B (MAO-B) inhibitors must be stable for at least 12 weeks prior to Screening.
* Levodopa administration at least 4 times daily (immediate or extended release) or three times daily (Rytary or Crexont).
* Stable use of oral anti-sialorrhea medications for 30 days before Screening, without anticipated need for change during the study.
* Average of ≥ 3 h total OFF time/day on Screening home diaries, with at least 2.5 hours OFF on each diary day.
* During Screening, capable of adequately identifying ON, OFF, and dyskinetic states (>80% concordance) through properly completed ON/OFF diaries.
* Female participants of childbearing potential and male participants with female partners of childbearing potential must agree to either remain abstinent or use adequate and reliable contraception throughout the study and for at least 12 weeks after the last dose of study drug has been taken.
* Able and willing to give written informed consent approved by an institutional review board, and to comply with scheduled visits, treatment plan, laboratory tests, and other study-related procedures.
* Approved as an appropriate and suitable candidate by the Enrollment Authorization Committee (EAC)

Exclusion Criteria:

* Diagnosis of secondary or atypical parkinsonism.
* Severe or disabling dyskinesias or OFF expected to preclude successful study participation, in the opinion of the investigator.
* Any previous procedure or therapy designed to provide continuous levodopa or stimulation of dopaminergic tone (i.e., Duopa, apomorphine, subcutaneous levodopa), surgery for PD (i.e., deep brain stimulation [DBS]), or anticipation of these during the study.
* History of exclusively diphasic, OFF state, myoclonic or dystonic dyskinesias without peak-dose choreiform dyskinesia.
* Clinically significant orthostatic hypotension (consistently symptomatic or requires medication).
* Clinically significant hallucinations requiring antipsychotic use.
* Current use of strong CYP3A4/5 inhibitors or inducers.
* Routine use of PD on-demand medications (i.e., inhaled levodopa, apomorphine injection). Routine use defined as three (3) or more uses per week of on-demand medication is not allowed. On demand medications should only be used for medical emergencies and should be avoided on anticipated diary days, as best as possible.
* Use of injectable botulinum medication for sialorrhea within 90 days of screening or during the study.
* Current use of medication with dopamine antagonist activity, or any use within 12 months of Screening.
* Clinically significant medical, surgical, psychiatric, or laboratory abnormalities that in the judgment of the investigator would preclude adequate participation or completion of the study.
* Clinically significant ECG abnormalities at Screening.
* Prolonged Fridericia-corrected QT (QTcF) interval on ECG at Screening.
* Clinically significant heart disease within 2 years of Screening, defined as follows:

  * Significant cardiac event within 12 weeks prior to Screening (e.g., admission for myocardial infarction, unstable angina, or decompensated heart failure), angina pectoris or episode of congestive heart failure with symptoms > grade 2 New York Heart Association classification, or presence of cardiac disease that in the opinion of the investigator increases the risk of ventricular arrhythmia.
  * History of complex arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia) that was symptomatic or required treatment.
  * Symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia
  * Symptomatic bradycardia, sick sinus syndrome or atrioventricular block greater than first degree in the absence of a pacemaker
  * Unexplained syncope
  * Brugada syndrome
  * Hypertrophic cardiomyopathy
* Any clinically significant history of malignancy or ongoing malignancy of sufficient concern for interference with completion of the study or quality of study experience, in the opinion of the investigator and medical monitor.
* Active major depressive disorder or a Beck Depression Inventory-II (BDI-II) score of > 19.
* Has active suicidal ideation within one year prior to Screening as determined by the C-SSRS or attempted suicide within the last 5 years.
* Has been diagnosed with or history of a substance-related disorder (excluding nicotine and caffeine), including alcohol-related disorder by Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria, during the 12 months prior to Screening.
* Tests positive at Screening for drugs of abuse. Drugs of abuse refers to illicit substances and does not include participants taking physician-prescribed medications. For participants who are legally prescribed cannabis for medical reasons, the appropriateness of the participant for this study will be made by the judgement of the Investigator in consultation with the Medical monitor.
* Has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than 2.5 times the upper limit of normal (ULN) or a degree of hepatic impairment using the Child-Pugh classification of B or C.
* Significant renal impairment as determined by estimated glomerular filtration rate (eGFR) less than or equal to 60 milliliters per minute (ml/min).
* Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCV) antibody, or Human Immunodeficiency Virus (HIV) infection at Screening.
* Currently lactating or pregnant or planning to become pregnant during the study.
* Previous exposure to CVN424.
* Currently participating in or has participated in another study of an investigational medicinal product (IMP) or medical device in the last 3 months or within 5 half-lives of the IMP (whichever is longer) prior to Screening.
* A known hypersensitivity to the IMP or to any excipients used in the formulation.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 12 in average daily OFF time on motor diaries for 150 mg CVN424 compared to placebo | Baseline and Up to Week 12
  The assessment of the average daily OFF time, normalized to waking hours will be based on diaries completed at home for three consecutive days during the 7-day period before a scheduled in-person visit.

SECONDARY OUTCOMES:
Change from Baseline to Week 12 in the ON time without troublesome dyskinesia | Baseline and Up to Week 12
  The assessment of the ON time without troublesome dyskinesia will be based on diaries completed at home for three consecutive days during the 7-day period before a scheduled in-person visit.
Change from Baseline to Week 12 on the Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II | Baseline and Up to Week 12
  The MDS-UPDRS is a comprehensive 50-question assessment of both motor and non-motor symptoms associated with PD. It features sections that require independent completion by people with PD and their caregivers, and sections to be completed by the same clinician throughout the study. Part II assess motor experiences of daily living, motor aspects of experiences of daily living. This part has 13 items. It is a self-administered questionnaire completed by the participant, which can be reviewed by the Investigator to ensure all responses are completed.
Change from Baseline to Week 12 on the Clinical Global Impression Scale - Severity (CGI-S) | Baseline and Up to Week 12
  The CGI-S is a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal/not at all ill) to 7 (amongst the most severely ill participants). This requires the clinician to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who have the same diagnosis. Higher scores indicate worser the illness.
Change from Baseline to Week 12 on the Patient Global Impression Scale - Severity (PGI-S) | Baseline and Up to Week 12
  The PGI-S is a participant-completed assessment rating PD severity on a scale of 1 to 5 with 1 being none and 5 being very severe. Higher scores indicate worser the illness.
Change from Baseline to Week 12 on the MDS-UPDRS Part III | Baseline and Up to Week 12
  The MDS-UPDRS is a comprehensive 50-question assessment of both motor and non-motor symptoms associated with PD. It features sections that require independent completion by people with PD and their caregivers, and sections to be completed by the same clinician throughout the study. Part III consists of 33 scores based on 18 items, and each question is anchored with five response scale from 0 (normal) to 4(severe). A 0 means there is no disability, and the higher the score, the more the disability is reflected. The maximum score for Part III is 132. The total score is the sum of the numerical response values of the items. It is completed by a rater based on findings from the motor examination.
Change from Baseline to Week 12 on the Epworth Sleepiness Scale (ESS) | Baseline and Up to Week 12
  The ESS is a participant self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0 to 3: would never doze, slight chance of dozing, moderate chance of dozing, and high chance of dozing), their usual chances of dozing off or falling asleep while engaged in eight different activities, such as sitting and reading, watching television, sitting in a public place, etc. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life, or their "daytime sleepiness". The questionnaire takes no more than 2 or 3 minutes to answer.
Change from Baseline to Week 12 in the ON time with no dyskinesia | Baseline and Up to Week 12
  The assessment of the ON time with no dyskinesia will be based on diaries completed at home for three consecutive days during the 7-day period before a scheduled in-person visit.
Change from Baseline to Week 12 on the MDS-UPDRS Part I | Baseline and Up to Week 12
  The MDS-UPDRS is a comprehensive 50-question assessment of both motor and non-motor symptoms associated with PD. It features sections that require independent completion by people with PD and their caregivers, and sections to be completed by the same clinician throughout the study. Part I assess non-motor experiences of daily living, non-motor aspects of experiences of daily living (6 items assessed by interview and 7 items by self-assessment). It has 13 items and is further grouped into two parts: Part IA has items associated with behaviors that are assessed and completed by the rater based on information provided by the participant and caregiver. Part IB is self-administered and completed by the participant with or without assistance or input from the caregiver, but independently of the rater. Responses to both IA and IB can be reviewed by the rater to ensure information accuracy and/or provide additional information or clarification of the test items, if necessary.
Change from Baseline to Week 12 on the Parkinson's Disease Questionnaire-39 (PDQ-39) | Baseline and Up to Week 12
  The PDQ is a 39-item self-report questionnaire that assesses eight PD-specific health related quality of life functions over the previous month. Assesses how often participants with PD experience difficulties across 8 dimensions of daily living including relationships, social situations and communication. The 39-item questionnaire offers a participant reported measure of health status and quality of life and is the most frequently used disease-specific health status measure. It also assesses the impact of PD on specific dimensions of functioning and wellbeing.
Change from Baseline to Week 12 on the Starkstein Apathy Scale (SAS) | Baseline and Up to Week 12
  The SAS instrument is used to identify apathy in participants with PD. The scale comprises 14 questions in which the respondent self-rates on a 4-point scale, ranging from "Not at all", "Slightly", "Some", and "A Lot". Ratings are a score from 3 to 0 for questions 1-8, and from 0 to 3 for questions 9-14, producing a total score out of 42. A score above 14 is considered the more severe level of apathy.
Change from Baseline to Week 12 on the CogState digital cognitive battery | Baseline and Up to Week 12
  Cogstate Digital Cognitive Testing Battery are computerized cognitive assessments of attention, executive function, verbal learning, and memory. It uses standardized scores to assess participant's cognitive function. These scores are transformed into a scale where the average performance of the general population is set at 100, with a standard deviation of 15. This means that a score of 100 represents average cognitive function, while scores above or below indicate better or poorer performance, respectively, compared to the average.
Change from Baseline to Week 12 on the Schwab and England (S & E) Activities of Daily Living Scale (ADL) | Baseline and Up to Week 12
  The Schwab and England Activities of Daily Living Scale is a commonly used tool to measure daily function for Parkinson's disease. The S & E Scale rates a PD participant's function on a scale from 0 indicating worst possible function to 100 indicating no impairment.
Number of participants reporting treatment emergent adverse events (TEAEs), TEAEs related to moderate or severe intensity and leading to withdrawal of study drug | Up to Week 14
Number of participants reporting serious adverse events (SAEs) | Up to Week 14
Number of participants with suicidal ideation as measured by Columbia Suicide Severity Rating Scale (C-SSRS) | Up to Week 12
Number of participants with impulse control disorders as measured by the Questionnaire for Impulsive-Compulsive Disorders in Parkinson 's disease Rating Scale (QUIP-RS) | Up to Week 12
  The QUIP-RS has 4 questions (common thoughts, urges/desires, self-control, faciliatory behaviors associated with impulse control disorders [ICDs]), each applied to 4 main impulse control disorders (gambling, buying, eating, and sexual behavior) and 3 related impulsivity disorders (medication use, punding, and hobbyism). Scores range from 0-4 for each question to gauge the frequency of behaviors over the preceding 4 weeks (or any defined 4-week period). Total scores range from 0 to 112.
Number of participants with clinically significant changes in physical examination, vital signs, electrocardiogram (ECG) finding, and laboratory values | Up to Week 14
Percentage of completers | Up to Week 12

OTHER OUTCOMES:
Maximum observed plasma concentration (Cmax) of CVN424 | At Day 1, Week 2, Week 4, Week 8, and Week 12
Time to reach Cmax of CVN424 | At Day 1, Week 2, Week 4, Week 8, and Week 12
Area under the plasma concentration-time curve from time 0 (time of dosing) to last time of sample collection hours (AUC 0-last) of CVN424 | At Day 1, Week 2, Week 4, Week 8, and Week 12
Half-life (t1/2) of CVN424 | At Day 1, Week 2, Week 4, Week 8, and Week 12
Change from Baseline on the Modality virtual assessments | Baseline and Up to Week 14
  The Modality System is an artificial intelligence interface designed to collect information on clinical performance through audio-visual conversational technology. Participants will engage with a virtual agent via a web browser on their electronic device, completing assessments aimed at testing various functions including speech, visuo-motor skills, prosodic (stress and intonation patterns), cognitive, and linguistic abilities.

CONTACTS AND LOCATIONS:
Locations (49):
- United States (45):
  - The Kirklin Clinic of UAB Hospital, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Parkinson's Research Centers of America - Orange county, Aliso Viejo, California
  - Parkinson's Research Centers of America - Palo Alto, Palo Alto, California
  - CenExel Rocky Mountain Clinical Research, Englewood, Colorado
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - SFM Clinical Research, LLC, Boca Raton, Florida
  - K2 Medical Research, Maitland, Florida
  - Renstar Medical Research, Ocala, Florida
  - N1 Research LLc, Orlando, Florida
  - Parkinson's Disease Center of SWFL, Port Charlotte, Florida
  - University Clinical Research-DeLand, LLC d/b/a Accel Research Sites - Brain & Spine Institute, Port Orange, Florida
  - USF Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Atlanta Neuroscience Institute, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Dept of Neurology Kentucky Neuroscience Institute Research, Lexington, Kentucky
  - Boston Clinical Trials, Boston, Massachusetts
  - University of Michigan Dept. of Neurology, Ann Arbor, Michigan
  - University of Michigan Hospital - Michigan Clinical Research Unit (MCRU), Ann Arbor, Michigan
  - Quest Research Institute, Farmington Hills, Michigan
  - Boro Neurology, Hopewell, New Jersey
  - Parkinson's Research Centers of America - Long Island, Commack, New York
  - Weill Cornell Medical College, New York, New York
  - The Neurological Institute, Charlotte, North Carolina
  - Duke Neurology Morreene Road Clinic, Durham, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Velocity Clinical Research, Raleigh, North Carolina
  - Riverhills Healthcare, Inc dba Riverhills Neuroscience, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Ohio State University - Martha Morehouse Medical Plaza, Columbus, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Veracity Neuroscience LLC, Memphis, Tennessee
  - Horizon Clinical Research Group, Cypress, Texas
  - Texas Movement Disorder Specialists, PLLC, Georgetown, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
  - Gill Neuroscience, Houston, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Inova Neurology - Fairfax, Fairfax, Virginia
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Henrico Doctors Neurology Associates, LLC, Richmond, Virginia
  - EvergreenHealth Research Department, Kirkland, Washington
  - Inland Northwest Research, Spokane, Washington
  - Medical College of Wisconsin-Department of Neurology, Milwaukee, Wisconsin
- Australia (3):
  - Southern Neurology, Kogarah, New South Wales
  - Westmead Hospital-Department of Neurology, Sydney, New South Wales
  - Perron Institute for Neurological and Translational Science, Nedlands, Western Australia
- The Alliance Hispanic Alliance for Clinical and Translational Research, Rio Piedras, Puerto Rico

IPD SHARING:
Plan to Share IPD: No